CLINICAL TRIAL: NCT01032174
Title: Non-Interventional Open Label Prospective Comparative Observational Study Of Evaluation Of Compliance In The Empiric Treatment With Azithromycin SR Versus Amoxiclav 1000 Mg In Adult Patients With Of Acute Bacterial Maxillary Sinusitis
Acronym: EASY
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0661199
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Maxillary Sinusitis
Keywords: Azithromycin SR Amoxiclav 1000 mg Maxillary Sinusitis
MeSH Terms: conditions — Maxillary Sinusitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Azithromycin SR: Acute Bacterial Maxillary Sinusitis
  Interventions: Drug: Azithromycin SR
- Amoxiclav 1000 mg: Acute Bacterial Maxillary Sinusitis
  Interventions: Drug: Amoxiclav 1000 mg

INTERVENTIONS:
Drug: Azithromycin SR — Azithromycin SR, 2.0 g by mouth (PO) x 1
  Groups: Azithromycin SR
Drug: Amoxiclav 1000 mg — Amoxiclav 1000 mg x twice daily, 10 days
  Groups: Amoxiclav 1000 mg

SUMMARY:
The purpose of this study is to compare compliance between patients with Acute Bacterial Sinusitis (ABS) treated with Azithromycin SR 2.0 g single dose orally and those treated with Amoxiclav - 1000 mg twice daily 10 days for the empiric treatment of ABS in outpatient clinic practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or nor pregnant or lactating female outpatients, 18 years of age or older.
* A clinical diagnosis of acute bacterial uncomplicated maxillary sinusitis as demonstrated by presence of the following signs and symptoms for a minimum duration of 7-10 days:

  1. Facial pain, pressure and/or tightness over one or both maxillary sinuses, and/or pain in one or both maxillary areas that worsens with movement or percussion, and
  2. Presence of one or more of the following signs:

  i.purulent nasal discharge ii.purulent drainage in the posterior pharynx iii.purulent discharge from the maxillary sinus orifice
* A sinus X-ray (Water's view) confirming the clinical diagnosis of maxillary sinusitis. At least one of the following must be documented in one or both maxillary sinuses on radiologic examination:

  1. complete or partial opacification
  2. an air/fluid level

Two or more of the following:

1. fever, as defined by temperature: >38ºC
2. leukocytosis [White Blood Cell (WBC) >10,000/mm3 or >15% band forms], ECR;
3. headache,
4. nasal congestion and post nasal drainage.

Exclusion Criteria:

* Known or suspected hypersensitivity or intolerance or contraindications to Azithromycin, Amoxiclav according to LPDs, pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Maxillary Sinusitis
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661199&StudyName=Non-Interventional%20Open%20Label%20Prospective%20Comparative%20Observational%20Study%20Of%20Evaluation%20Of%20Compliance%20In%20The%20Empiric%20Treatment%20With%20Azithromyc

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: A single dose of azithromycin 2000 milligram (mg) sustained release (SR) tablet administered orally.
- Amoxiclav: Amoxiclav 1000 mg tablet administered twice daily (BID) orally for 10 days.
Period: Overall Study
Arm/Group | Azithromycin | Amoxiclav
Started | 63 | 60
Completed | 63 | 59
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Amoxiclav | Total
Number analyzed (Participants) | 63 | 60 | 123
Age Continuous [Mean (Standard Deviation); unit: years] | 36.9 (11.6) | 38.4 (13.4) | 37.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 34 | 64
  Male | 33 | 26 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response of Very Convenient or Somewhat Convenient
Description: Participant reported outcome questionnaire was the assessment of participant's convenience with drug treatment based on following categories: very convenient or somewhat convenient and not convenient or not at all convenient. Value of 1 was reported if participant answered 'very convenient' or 'somewhat convenient' and 0 if participant answered 'not convenient' or 'not at all convenient'.
Time Frame: Day 11
Population: The Full Analysis Set (FAS) population included all participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy evaluation. 'N' signifies number of participants with non-missing data. Missing observations were not imputed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Azithromycin | Amoxiclav
Number analyzed (Participants) | 63 | 59
Percentage of Participants | 100.0 | 72.9
Statistical Analysis 1: Comparison: Azithromycin vs Amoxiclav; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — The logistic regression model contained terms for treatment, gender and age

2. Secondary Outcome: Percent Compliance With Prescribed Treatment Regimen
Description: Percent compliance with the prescribed treatment regimen was calculated as 100 multiplied by (number of tablets taken by the participant divided by number of tablets prescribed).
Time Frame: Day 11
Population: The FAS population included all participants who received at least 1 dose of study medication and had at least 1 post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: Percent compliance
Arm/Group | Azithromycin | Amoxiclav
Number analyzed (Participants) | 63 | 60
Percent compliance | 100.00 (0.00) | 99.00 (3.88)
Statistical Analysis 1: Comparison: Azithromycin vs Amoxiclav; Test type: Superiority or Other; p = 0.0568, ANCOVA — The analysis of covariance (ANCOVA) model contained terms for treatment, gender, age and Body Mass Index (BMI); Least square mean was adjusted for gender, age and BMI; Difference of Least Square Mean = 1.06, 95% CI 2-sided [-0.03 to 2.15], Standard Error of Mean 0.55

3. Secondary Outcome: Percentage of Participants Who Were 100 Percent Compliant With Prescribed Treatment Regimen
Description: Percent compliance with the prescribed treatment regimen was calculated as 100 multiplied by (number of tablets taken by the participant divided by number of tablets prescribed). Value of 1 was reported if percent compliance equals to 100, and 0 if percent compliance was non-missing and less than 100.
Time Frame: Day 11
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Azithromycin | Amoxiclav
Number analyzed (Participants) | 63 | 60
Percentage of Participants | 100.0 | 91.7
Statistical Analysis 1: Comparison: Azithromycin vs Amoxiclav; Test type: Superiority or Other; p = 0.0682, Regression, Logistic — The logistic regression model contained terms for treatment, gender and age

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Azithromycin | Amoxiclav
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/60
Other Adverse Events (participants affected / at risk) | 7/63 | 9/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=63) | Amoxiclav (N=60)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 2
Vulvovaginal candidiasis (Infections and infestations) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.